CLINICAL TRIAL: NCT04501016
Title: A Stepped Care Approach to Treating Tobacco Use in Rural Veterans
Acronym: Stepped Care
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Iowa City Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mark Vander Weg, Core Investigator, Iowa City Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IowacityVAMC
Record Dates: First submitted 2020-07-29; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Tobacco Cessation
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Intervention Model Description: All tobacco users will receive a tailored pharmacological and behavioral intervention. The specific counseling protocol will vary depending upon their response to treatment and initial success with quitting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tailored Intervention (Experimental): Tailored behavioral counseling combined with tobacco cessation pharmacotherapy.
  Interventions: Behavioral: Tailored behavioral counseling; Drug: Tobacco cessation pharmacotherapy

INTERVENTIONS:
Behavioral: Tailored behavioral counseling — Participants will initially receive a six-session telephone intervention. Standard cognitive behavioral treatment strategies will be included. Participants will be screened for elevated depressive symptoms, risky alcohol use, and concerns about weight and and offered supplemental behavioral counseling related to these issues as appropriate. Those that are unable to quit tobacco initially will receive an enhanced, four-session counseling module focused on reduced scheduled smoking. Those who do quit tobacco use initially will receive four sessions of extended counseling based on positive psychology intervention strategies.
Drug: Tobacco cessation pharmacotherapy — Pharmacotherapy will be selected based on medical and psychiatric history and potential interactions with other current medications combined with shared decision making. Options will include nicotine gum (2 and 4 mg), nicotine lozenge (2 and 4 mg), nicotine patch (7, 14, and 21 mg), bupropion (150 mg twice daily) and varenicline (1 mg twice daily). Monotherapy and combination therapy options will be provided.

SUMMARY:
Tobacco use remains prevalent among Veterans. Although effective smoking cessation interventions exist, long-term term quit rates remain sub-optimal. The project will investigate the feasibility of a stepped care approach to treating tobacco use that includes enhancements based on initial response to treatment to augment the investigators' existing tailored tobacco treatment intervention.

DETAILED DESCRIPTION:
Rural tobacco users (cigarette smokers, smokeless tobacco users, and users of other forms of tobacco) from the Iowa City VA Health Care System will be proactively recruited using information obtained from the electronic medical record. All participants will receive the investigators' tailored, six session smoking cessation intervention developed over a series of projects funded by ORH. This includes a counseling protocol tailored to tobacco users' individual needs and associated risk factors as well as pharmacotherapy selected using shared decision making. Participants who are unable to quit initially will be provided with enhanced counseling based on self-monitoring and scheduled reduced smoking. Those who are able to quit using tobacco during the initial treatment phase will be given an extended, four-session counseling protocol that incorporates new content based on established interventions from positive psychology in an effort to reduce relapse.

ELIGIBILITY:
Inclusion Criteria:

* Use tobacco (cigarettes, smokeless tobacco, pipes, cigars, hookah) on a daily basis
* Be willing to make a quit attempt in the next 30 days
* Able to provide informed consent
* Have access to a telephone
* Have a stable residence,

Exclusion Criteria:

* Planning to move within the next 6 months
* Terminal illness
* Unstable psychiatric disorder (e.g., acute psychosis)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Tobacco cessation | 6 months
  7-day point prevalence tobacco cessation

SECONDARY OUTCOMES:
Tobacco cessation | 3 months
  7-day point prevalence tobacco cessation
Salivary cotinine levels (in ng/ml) | 6 months
  Salivary cotinine

OTHER OUTCOMES:
Level of satisfaction with the intervention as measured according to a five-point scale (extremely, very, moderately, slightly, not at all) | 3 months
  Self-reported satisfaction with the intervention according to the dimensions of usefulness, convenience, difficulty, liking, and helpfulness using five response options (extremely, very, moderately, slightly, not at all) using a scale developed specifically for the project.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Vander Weg, PhD, Principal Investigator — Iowa City VA Health Care System
Locations (1):
- Iowa City VA Healthcare System, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No